CLINICAL TRIAL: NCT04628910
Title: Examining the Differential Effects of Traditional Float-REST and Dry Float on Subjective and Objective Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2006024602
Record Dates: First submitted 2020-09-24; First posted 2020-11-16 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-04

CONDITIONS: Sleep Quality
Keywords: Sleep; Sensory Deprivation Tank; Wearable Technology; Dry Float
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Weeks 0-1: Testing battery; begin daily surveys and at home monitoring via smartphone applications. This will serve as baseline and will be collected for, at minimum, 5 days prior to the first experimental condition.
  Weeks 2-4: Complete daily surveys and at home monitoring via smartphone applications; Complete the first experimental condition (Float-REST or Dry Float) in 60 minute sessions, twice a week.
  Week 5: Complete daily surveys and at home monitoring via smartphone applications. A second round of the testing battery will be completed prior to beginning the next condition.
  Week 6-8: Complete daily surveys and at home monitoring via smartphone applications; Complete the first experimental condition (Float-REST or Dry Float) in 60 minute sessions, twice a week.
  Week 9: Complete daily surveys and at home monitoring via smartphone applications. The testing battery will be completed for the final time toward the end of the week and will signify their completion of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Float-REST Therapy (Active Comparator): Participants will utilize sensory deprivation tanks.
  Interventions: Other: Traditional Float-REST Therapy
- Simulated Flotation Therapy (Experimental): Participants will utilize the Zerobody dry flotation therapy.
  Interventions: Other: Simulated Flotation Therapy

INTERVENTIONS:
Other: Simulated Flotation Therapy — The Zerobody is a new technology designed to simulate the effects of traditional Float-REST therapy, but without the contact with salt water. The system has a very thin membrane that cradles the body and provides a warm sensation, similar to that experienced in a traditional flotation tank. The system will be housed in a room that allows for significant reductions in light and sound to mimic the experience of a flotation tank. The room will contain an intercom that allows participants to communicate with study personnel in the event they need assistance. Participants will undergo 60 minute sessions twice a week for 3 weeks using the Zerobody, also termed "dry floating," as one of the two interventions.
  Other Names: Zerobody Dry Float
  Arms: Simulated Flotation Therapy
Other: Traditional Float-REST Therapy — Traditional Float-REST therapy uses sensory deprivation tanks that consist of a very large warm water enclosure with a high concentration of Epsom salt to create a completely buoyant environment. This, along with a combination of temperature that is kept equal to skin temperature (94 degrees), allows the participant to eliminate the gravitational effects on the body, and along with lack of sound and low to no light (depending on comfort) allows the brain and body to completely relax for augmented physical and mental recovery. The room will contain an intercom that allows participants to communicate with study personnel in the event they need assistance. Participants will undergo 60 minute sessions twice a week for 3 weeks as one of the two interventions.
  Other Names: Sensory Deprivation Tanks
  Arms: Traditional Float-REST Therapy

SUMMARY:
The objective of this research study is to assess how the implementation of various modern strategies for augmented recovery affect sleep quality, subjective wellness and other indices of general well-being.

DETAILED DESCRIPTION:
Traditional flotation therapy (Float-REST; Flotation Restricted Environmental Stimulation Therapy) uses sensory deprivation tanks that consist of a very large warm water enclosure with a high concentration of Epsom salt to create a completely buoyant environment. This, along with a combination of temperature that is kept equal to skin temperature (94 degrees), allows the participant to eliminate the gravitational effects on the body, and along with lack of sound and low to no light (depending on comfort) allows the brain and body to completely relax for augmented physical and mental recovery. Provided the growing understanding that sleep quality and quantity are at the forefront of ensuring optimal human performance states, compounded by the deleterious effects of high stress and anxiety on sleep, utilizing flotation therapy as a mechanism for enhancing sleep requires further investigation. In addition to the traditional Float- REST, there have been developments in newer technologies that enhance the convenience of receiving these proposed benefits; Zerobody Dry Float technology (www.Zerobody.com) rids the need for multiple showers by its user, frequent water treatments, and extensive maintenance experienced with traditional flotation environments. However, research is still needed to assess how this recovery modality compares to traditional Float-REST.

To assess whether traditional (Float-REST) or simulated (Dry Float) flotation therapy positively influences sleep and perceptual recovery, participants will undergo a crossover study. Over the course of 9 weeks, participants will alternate Float-REST and Dry Float in 3 week segments with a 1 week break in-between to gather baseline data (known as the testing battery). In addition, testing battery data will be collected at weeks 1 and 9. The order in which participants begin their crossover study, either Float-REST or Dry Float, will be randomly assigned. All participants may wear a fitness tracker and a sleep monitoring ring worn on the finger for the duration of the study. In addition, daily, per session, and pre/post-study questionnaires will be submitted via a smartphone application.

ELIGIBILITY:
Inclusion Criteria:

• Male or female 18-60 years of age

Exclusion Criteria:

* Weighs more than 250 pounds
* Taller than 76 inches
* Has undergone a float-REST session of any kind in the last 3 months
* Has a fresh piercings that is less than 6 weeks old from scheduled session
* Has a fresh tattoo that is less than 4 weeks old from scheduled float
* Has an injury requiring an orthopedic cast (i.e. plaster or synthetic), immovable splint or brace
* Is claustrophobic (fear of confined spaces)
* Has a skin or respiratory sensitivity or allergy to chlorine, sulfate, magnesium, rubber latex or synthetic latex
* Has a history of or is prone to motion sickness
* Has had an episode of loss of consciousness in the last 6-months
* Has had a concussion or traumatic brain injury in the last 6-months
* Has a contagious skin conditions
* Has skin ulcers, open rashes, incisions, stitches or large open wounds that could cause pain when exposed to saltwater
* Has a diagnosis of kidney disease, heart disease or other chronic illness
* Has a irremovable medical port or catheter
* Has had a seizure in the last 10 years
* Has communicable diseases (e.g. HIV, Hepatitis A, B & C, tuberculosis, or measles)
* Lack of control of bodily functions prior to scheduled float
* Has a diagnosis of any psychiatric condition (e.g. schizophrenia or bipolar disorder)
* Pregnant or actively trying to become pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-04-17 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Change in heart rate variability as measured by OURA ring | Daily from baseline through study completion at 9 weeks
  Oura Ring is a connected health device worn on the finger that measures sleep. Heart rate variability will be quantified throughout the night via the OURA ring.
Change in heart rate as measured by OURA ring | Daily from baseline through study completion at 9 weeks
  Oura Ring is a connected health device worn on the finger that measures sleep. Heart rate will be quantified throughout the night via the OURA ring.
Change in per session self-report measures | 2 times a week, in 3 week increments, through study completion at 9 weeks
  State-Trait Anxiety Index (STAI) - Commonly used measure of state and trait anxiety, and done with 20 very brief questions. Values range from 20 to 80, with higher scores representing more severe anxiety. Participants will complete the STAI questionnaire before and after each session, twice a week. The sessions will take place during weeks 2-4 and weeks 6-8.
Change in testing battery self-report measures in sleep quality | Week 1, week 5, and week 9
  Pittsburgh Sleep Quality Index (PSQI)- 19 item inventory with 7 subjective components that assess sleep quality over time. Each component is scored from 0 to 3 (0=very good and 3=very bad). The sum of the components is the global score and ranges 0-21 (0=no difficulty and 21=severe difficulties). The higher the global score, the poorer the sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Rockefeller Neuroscience Institute at West Virginia University, Morgantown, West Virginia, United States